CLINICAL TRIAL: NCT01595295
Title: Registry on Hypomethylating Agents in Myeloid Neoplasms, Including Myelodysplastic Syndromes (MDS), Chronic Myelomonocytic Leukemia (CMML) and Acute Myeloid Leukemia (AML)
Brief Title: Registry on Hypomethylating Agents in Myeloid Neoplasms
Status: Completed | Type: Observational
Sponsor: Arbeitsgemeinschaft medikamentoese Tumortherapie (Other)
Responsible Party: Sponsor
Other Study IDs: AGMT_HMA Register
Record Dates: First submitted 2012-05-07; First posted 2012-05-10 (Estimated); Last update posted 2024-03-25 (Actual); Status verified 2024-03

CONDITIONS: Chronic Myelomonocytic Leukemia; Myelodysplastic Syndromes; Acute Myeloid Leukemia
Keywords: CMML; MDS; AML; registry; Vidaza
MeSH Terms: conditions — Leukemia, Myelomonocytic, Chronic; Myelodysplastic Syndromes; Leukemia, Myeloid, Acute

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples With DNA — From some patients with myeloid neoplasms blood or tissue samples will be stored for further analyses. These samples will also be obtained from patients, who are not or not yet treated with hypomethylating agents, to comprise a control.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Hypomethylating Agents: Patients treated with hypomethylating agents
  Interventions: Other: non interventional

INTERVENTIONS:
Other: non interventional

SUMMARY:
This registry is set up to collect real-world experience in the management of patients with myeloid neoplasms, in particularly in patients with MDS, CMML or AML, treated with hypomethylating agents in Austria and potentially other participating countries. This registry will collect data in a retrospective as well as in a prospective manner at various sites. The aim is to gain valuable insights on both efficacy and toxicity of these drugs in a routine clinical setting in patients with various comorbidities.

ELIGIBILITY:
Inclusion Criteria:

Patients with MDS, CMML, and AML

* who begin with or already have received treatment with with a hypomethylating agent
* who are willing to provide informed consent

Exclusion Criteria:

* Due to the non-interventional design of this program there are no specific exclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with MDS, CMML, and AML, who begin with or already have received treatment with a hypomethylating agent
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Actual)
Dates: Start 2009-02-09 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Response evaluation | up to 10 years
  hematological response, marrow response, cytogenetic response (if data is available), quantification of reduced need for transfusions, median response duration
Overall survival | up to 10 years

SECONDARY OUTCOMES:
Documentation of adverse events and toxicities | up to 10 years
Number of treatment cycles | up to 10 years
Number and reasons of dose reductions | up to 10 years
Uni/multivariate analysis of various factors known or thought to influence overall survival in order to establish prognostic markers | up to 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Richard Greil, MD, Study Chair — Universitätsklinik für Innere Medizin III der PMU Salzburg; Lisa Pleyer, MD, Principal Investigator — Universitätsklinik für Innere Medizin III der PMU Salzburg
Locations (20):
- Austria (19):
  - LKH Feldkirch, Innere Med. II, Interne E, Feldkirch
  - LKH Fürstenfeld, Fürstenfeld
  - UK Graz: Universitätsklinik für Innere Medizin; Klinische Abteilung für Hämatologie, Graz
  - Universitätsklinik für Innere Medizin V, Innsbruck
  - Klinikum Klagenfurt: 1. Medizinische Abteilung, Klagenfurt
  - UK Krems: Innere Medizin II, Krems
  - LKH Hochsteiermark, Leoben
  - Ordensklinikum Linz - BHS: Interne I: Medizinische Onkologie und Hämatologie, Linz
  - Ordensklinikum Linz - Elisabethinen: Interne I, Linz
  - Kepler Universitätsklinikum Linz, Med. Campus III., Univ.-Klinik für Hämatologie und Internistische Onkologie, Linz
  - Universitätsklinik für Innere Medizin III Universitätsklinik für Innere Medizin III der PMU Salzburg, Salzburg
  - Klinikum Steyr: Innere Medizin II: Onkologie, Gastroenterologie, Angiologie, Steyr
  - Klinik Landstraße: 1. Medizinische Abteilung, Vienna
  - AKH Meduni Wien: Universitätsklinik für Innere Medizin I: Klinische Abteilung für Hämatologie und Hämostaseologie, Vienna
  - Krankenhaus Hietzing, Vienna
  - Hanusch Krankenhaus, Vienna
  - Klinik Ottakring, 1. Med. Abteilung, Vienna
  - Klinik Donaustadt: 2. Medizinische Abteilung, Vienna
  - Klinikum Wels Grieskirchen, Wels
- Clinical Hospital Merkur, Zagreb, Croatia

REFERENCES:
- [Result] Pleyer L, Stauder R, Burgstaller S, Schreder M, Tinchon C, Pfeilstocker M, Steinkirchner S, Melchardt T, Mitrovic M, Girschikofsky M, Lang A, Krippl P, Sliwa T, Egle A, Linkesch W, Voskova D, Angermann H, Greil R. Azacitidine in patients with WHO-defined AML - results of 155 patients from the Austrian Azacitidine Registry of the AGMT-Study Group. J Hematol Oncol. 2013 Apr 29;6:32. doi: 10.1186/1756-8722-6-32. PMID 23627920
- [Result] Pleyer L, Burgstaller S, Girschikofsky M, Linkesch W, Stauder R, Pfeilstocker M, Schreder M, Tinchon C, Sliwa T, Lang A, Sperr WR, Krippl P, Geissler D, Voskova D, Schlick K, Thaler J, Machherndl-Spandl S, Theiler G, Eckmullner O, Greil R. Azacitidine in 302 patients with WHO-defined acute myeloid leukemia: results from the Austrian Azacitidine Registry of the AGMT-Study Group. Ann Hematol. 2014 Nov;93(11):1825-38. doi: 10.1007/s00277-014-2126-9. Epub 2014 Jun 21. PMID 24951123
- [Result] Pleyer L, Germing U, Sperr WR, Linkesch W, Burgstaller S, Stauder R, Girschikofsky M, Schreder M, Pfeilstocker M, Lang A, Sliwa T, Geissler D, Schlick K, Placher-Sorko G, Theiler G, Thaler J, Mitrovic M, Neureiter D, Valent P, Greil R. Azacitidine in CMML: matched-pair analyses of daily-life patients reveal modest effects on clinical course and survival. Leuk Res. 2014 Apr;38(4):475-83. doi: 10.1016/j.leukres.2014.01.006. Epub 2014 Jan 18. PMID 24522248
- [Result] Ramos F, Thepot S, Pleyer L, Maurillo L, Itzykson R, Bargay J, Stauder R, Venditti A, Seegers V, Martinez-Robles V, Burgstaller S, Recher C, Deben G, Gaidano G, Gardin C, Musto P, Greil R, Sanchez-Guijo F, Fenaux P; European ALMA Investigators. Azacitidine frontline therapy for unfit acute myeloid leukemia patients: clinical use and outcome prediction. Leuk Res. 2015 Mar;39(3):296-306. doi: 10.1016/j.leukres.2014.12.013. Epub 2014 Dec 31. PMID 25601157
- [Result] Pleyer L, Burgstaller S, Stauder R, Girschikofsky M, Sill H, Schlick K, Thaler J, Halter B, Machherndl-Spandl S, Zebisch A, Pichler A, Pfeilstocker M, Autzinger EM, Lang A, Geissler K, Voskova D, Geissler D, Sperr WR, Hojas S, Rogulj IM, Andel J, Greil R. Azacitidine front-line in 339 patients with myelodysplastic syndromes and acute myeloid leukaemia: comparison of French-American-British and World Health Organization classifications. J Hematol Oncol. 2016 Apr 16;9:39. doi: 10.1186/s13045-016-0263-4. PMID 27084507
- [Result] Pleyer L, Dohner H, Dombret H, Seymour JF, Schuh AC, Beach CL, Swern AS, Burgstaller S, Stauder R, Girschikofsky M, Sill H, Schlick K, Thaler J, Halter B, Machherndl Spandl S, Zebisch A, Pichler A, Pfeilstocker M, Autzinger EM, Lang A, Geissler K, Voskova D, Sperr WR, Hojas S, Rogulj IM, Andel J, Greil R. Azacitidine for Front-Line Therapy of Patients with AML: Reproducible Efficacy Established by Direct Comparison of International Phase 3 Trial Data with Registry Data from the Austrian Azacitidine Registry of the AGMT Study Group. Int J Mol Sci. 2017 Feb 15;18(2):415. doi: 10.3390/ijms18020415. PMID 28212292
- [Result] Almeida AM, Prebet T, Itzykson R, Ramos F, Al-Ali H, Shammo J, Pinto R, Maurillo L, Wetzel J, Musto P, Van De Loosdrecht AA, Costa MJ, Esteves S, Burgstaller S, Stauder R, Autzinger EM, Lang A, Krippl P, Geissler D, Falantes JF, Pedro C, Bargay J, Deben G, Garrido A, Bonanad S, Diez-Campelo M, Thepot S, Ades L, Sperr WR, Valent P, Fenaux P, Sekeres MA, Greil R, Pleyer L. Clinical Outcomes of 217 Patients with Acute Erythroleukemia According to Treatment Type and Line: A Retrospective Multinational Study. Int J Mol Sci. 2017 Apr 14;18(4):837. doi: 10.3390/ijms18040837. PMID 28420120
- [Result] Leisch M, Weiss L, Lindlbauer N, Jungbauer C, Egle A, Rohde E, Greil R, Grabmer C, Pleyer L. Red blood cell alloimmunization in 184 patients with myeloid neoplasms treated with azacitidine - A retrospective single center experience. Leuk Res. 2017 Aug;59:12-19. doi: 10.1016/j.leukres.2017.05.006. Epub 2017 May 9. PMID 28535394
- [Result] Huemer F, Weiss L, Faber V, Neureiter D, Egle A, Geissler K, Voskova D, Zebisch A, Burgstaller S, Pichler A, Stauder R, Sperr W, Lang A, Pfeilstocker M, Machherndl-Spandl S, Stampfl M, Greil R, Pleyer L. Establishment and validation of a novel risk model for estimating time to first treatment in 120 patients with chronic myelomonocytic leukaemia. Wien Klin Wochenschr. 2018 Feb;130(3-4):115-125. doi: 10.1007/s00508-018-1315-2. Epub 2018 Jan 30. PMID 29383443
- [Result] Falantes J, Pleyer L, Thepot S, Almeida AM, Maurillo L, Martinez-Robles V, Stauder R, Itzykson R, Pinto R, Venditti A, Bargay J, Burgstaller S, Martinez MP, Seegers V, Cortesao E, Foncillas MA, Gardin C, Montesinos P, Musto P, Fenaux P, Greil R, Sanz MA, Ramos F; European ALMA + Investigators. Real life experience with frontline azacitidine in a large series of older adults with acute myeloid leukemia stratified by MRC/LRF score: results from the expanded international E-ALMA series (E-ALMA+). Leuk Lymphoma. 2018 May;59(5):1113-1120. doi: 10.1080/10428194.2017.1365854. Epub 2017 Aug 24. PMID 28838276
- [Result] Pleyer L, Leisch M, Kourakli A, Padron E, Maciejewski JP, Xicoy Cirici B, Kaivers J, Ungerstedt J, Heibl S, Patiou P, Hunter AM, Mora E, Geissler K, Dimou M, Jimenez Lorenzo MJ, Melchardt T, Egle A, Viniou AN, Patel BJ, Arnan M, Valent P, Roubakis C, Bernal Del Castillo T, Galanopoulos A, Calabuig Munoz M, Bonadies N, Medina de Almeida A, Cermak J, Jerez A, Montoro MJ, Cortes A, Avendano Pita A, Lopez Andrade B, Hellstroem-Lindberg E, Germing U, Sekeres MA, List AF, Symeonidis A, Sanz GF, Larcher-Senn J, Greil R. Outcomes of patients with chronic myelomonocytic leukaemia treated with non-curative therapies: a retrospective cohort study. Lancet Haematol. 2021 Feb;8(2):e135-e148. doi: 10.1016/S2352-3026(20)30374-4. PMID 33513373
- [Result] Leisch M, Pfeilstocker M, Stauder R, Heibl S, Sill H, Girschikofsky M, Stampfl-Mattersberger M, Tinchon C, Hartmann B, Petzer A, Schreder M, Kiesl D, Vallet S, Egle A, Melchardt T, Piringer G, Zebisch A, Machherndl-Spandl S, Wolf D, Keil F, Drost M, Greil R, Pleyer L. Adverse Events in 1406 Patients Receiving 13,780 Cycles of Azacitidine within the Austrian Registry of Hypomethylating Agents-A Prospective Cohort Study of the AGMT Study-Group. Cancers (Basel). 2022 May 17;14(10):2459. doi: 10.3390/cancers14102459. PMID 35626063
- [Result] Pleyer L, Sekeres MA. An early glimpse at azacitidine plus venetoclax for myelodysplastic syndromes. Lancet Haematol. 2022 Oct;9(10):e714-e716. doi: 10.1016/S2352-3026(22)00252-6. Epub 2022 Sep 2. No abstract available. PMID 36063831